CLINICAL TRIAL: NCT01086852
Title: A Phase III Open, Multicentre Study to Investigate the Safety and Efficacy of BPL's High Purity FACTOR X in the Treatment of Factor X Deficient Subjects Undergoing Surgery
Brief Title: Safety & Efficacy of BPL's High Purity FACTOR X in Treatment of Factor X Deficient Subjects Undergoing Surgery
Acronym: Ten03
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed early due to difficulties in enrolling the target number of 10 surgical procedures.
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ten03
Record Dates: First submitted 2009-11-10; First posted 2010-03-15 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Factor X Deficiency
Keywords: Factor X deficiency; surgery; Factor X deficiency subjects requiring surgery
MeSH Terms: conditions — Factor X Deficiency | interventions — Factor X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FACTOR X (Experimental): Human Coagulation Factor X
  Interventions: Biological: FACTOR X

INTERVENTIONS:
Biological: FACTOR X — Presurgery loading dose- The FX level of 70%-90% should be achieved.This will be calculated based on the patients weight on day of surgery and the required rise. Initial dose should not exceed 60IU/kg.
  Post surgery- FX trough levels of 50% should be achieved.
  Intravenous infusion of factor X is given at a suggested rate of 10mL/min but not exceeding more than 20mL/min.

SUMMARY:
To primary efficacy variable is to assess the presence or absence of excessive blood loss during and after surgery.

The secondary efficacy endpoints are as follows:

1. A subjective overall assessment by the investigator of FACTOR X in the control of bleeding during surgery.
2. The incidence of bleeding episodes during treatment with FACTOR X while the subject is at risk of post-operative bleeding, including location and duration.
3. Incremental recovery of FX:C and FX:Ag after the pre-surgery bolus infusion.
4. Assessment of FX:C and FX:Ag levels on each day post-surgery.
5. Assessment of the cumulative weight-adjusted doses of FACTOR X as measured by FX:C (IU/kg body weight) administered to each subject to maintain haemostasis.
6. Assessment of the cumulative doses of FACTOR X as measured by FX:C (IU) administered to each subject to maintain haemostasis.
7. Amount of weight-adjusted FACTOR X as measured by FX:C (IU/kg body weight) administered daily (day of surgery and each post-operative day) to maintain haemostasis.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of FACTOR X administered by bolus infusion to prevent bleeding and achieve haemostasis in factor X deficient subjects undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 12 years of age at date of written informed consent/assent.
* Subjects who have given written informed consent or, for subjects aged 12-17 years (inclusive), have given written assent and whose parent/guardian has given written informed consent.
* Subjects with hereditary mild to severe Factor X deficiency (<20% basal FX activity), including previously untreated subjects OR those currently treated with Fresh Frozen Plasma (FFP), Prothrombin Complex Concentrate (PCC) or factor IX/X concentrate by prophylaxis or on demand.
* Subjects who are to undergo surgery in which the investigator believes a factor X concentrate will be required due to a prior history of unusual bleeding either spontaneously or after surgery or trauma in the absence of treatment with a factor X containing product.
* Pregnant subjects undergoing obstetric delivery (including Caesarean surgery and vaginal delivery) may enter the study. Female subjects of child-bearing potential must have a negative result on a human chorionic gonadotropin-based pregnancy test. If a female subject is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study.

Exclusion Criteria:

* Subjects who are required or expected to take other factor X containing medications during or after surgery.
* Subjects with a history of inhibitor development to FX or a detectable inhibitor to FX (≥0.6 BU) on the Nijmegen-Bethesda assay at screening. Obtaining a FX inhibitor result at screening is not mandatory if the subject is to undergo emergency surgery and the local laboratory is unable to perform the analyses prior to the surgical procedure.
* Subjects with thrombocytopenia (platelets < 50 x 109/L).
* Subjects who have clinically significant renal disease (creatinine >200µmol/L).
* Subjects who have clinically significant liver disease (ALT levels greater than three times the upper limit of normal).
* Subjects known to have other coagulopathy or thrombophilia.
* Subjects who are currently participating or have participated in another trial within the last 30 days, with the exception of the BPL Factor X PK study (protocol number Ten01).
* Female subjects who are lactating.
* Subjects who have known or suspected hypersensitivity to the investigational medicinal product or its excipients.
* Subjects known to have abused chemicals or drugs within the past 12 months.
* Subjects with a history of unreliability or non-cooperation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Aldwinckle, Principal Investigator — Bio Products Laboratory
Locations (7):
- University Of Texas Health Science Center, Gulf States Hemophilia and Thrombophilia Center 6655 Travis St, Houston, Texas, United States
- Unidad Coagulopatías, Congenitas, Edificio Dotacional, 1ra Planta Hospital Universito La Paz, Madrid, Spain
- Turkey (Türkiye) (2):
  - Ege University School of Medicine, Departmant of Pediatric Hematology, Bornova, İzmir
  - Istanbul University Cerrahpasa Medicine Faculty Department of Pediatric Hematology, Istanbul
- United Kingdom (3):
  - Department of Hematology, Royal Cornwall Hospital,, Truro, Cornwall
  - The Katherine Dormandy Haemophilia Centre and Thrombosis Unit, The Royal Free Hospital,Pond Street, Hampstead, London
  - Hammersmith Hospital, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment With FACTOR X: Four subjects underwent 4 major surgeries with active treatment (FACTOR X)
Period: Overall Study
Arm/Group | Active Treatment With FACTOR X
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment With FACTOR X: Four patients underwent 4 major surgeries with active treatment (FACTOR X)
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [55 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
  United Kingdom | 2
FX:C at diagnosis (IU/dL) [Median (Full Range); unit: IU/dL] | 7.5 [7 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Estimation of Volume of Blood Loss During Surgery
Description: As soon as possible after wound closure, the investigator estimated the volume of blood loss during surgery and made a clinical assessment against the volume of blood loss typically expected in a normal patient (i.e. one without a bleeding disorder and undergoing the same surgical procedure). The assessment may have been supported by a swab and pad count.
  The clinical assessment was rated as follows:
  * Blood loss less than expected
  * Blood loss as expected
  * Blood loss more than expected
  * Blood loss excessive (defined as more than twice the pre defined amount that would be expected in a normal patient for this type of surgery)
Time Frame: Blood loss is measured during and after surgery, the overall assessment is made after the last dose of FACTOR X.
Population: The ITT population will be defined as all surgical procedures in which subjects were treated with at least one dose of FACTOR X and have undergone surgery.
Measure: Geometric Mean (Standard Deviation); unit: ml
Groups:
- FACTOR X: Human Coagulation Factor X
  FACTOR X: Presurgery loading dose- The FX level of 70%-90% should be achieved.This will be calculated based on the patients weight on day of surgery and the required rise. Initial dose should not exceed 60IU/kg.
  Post surgery- FX trough levels of 50% should be achieved.
  Intravenous infusion of factor X is given at a suggested rate of 10mL/min but not exceeding more than 20mL/min.
Arm/Group | FACTOR X
Number analyzed (Participants) | 4
ml | 160.5 (168.49)

2. Secondary Outcome: Incremental Recovery After Bolus Dose of FACTOR X
Description: Incremental Recovery of FX:C after the Pre surgery Bolus Infusion The factor X increment is calculated by subtracting the pre-infusion factor X level from the post-dose value.
  Incremental recovery is calculated by FX increment (IU/dL)/ FX dose (IU/kg)
Time Frame: incremental recovery was assessed at approximately 30 minutes after the pre surgery bolus
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | FACTOR X
Number analyzed (Participants) | 4
IU/dL per IU/kg | 2.14 (0.224)

3. Primary Outcome: Clinical Assessment of Blood Loss During Surgery Against the Volume of Blood Loss Expected in Patients Without a Bleeding Disorder.
Description: The investigator's estimation of the volume of blood loss during surgery compared to the volume of blood loss expected in patients without a bleeding disorder undergoing the same surgical procedure and reported as greater than, equal to or less than.
Time Frame: After wound closure
Population: All subjects treated with FACTOR X
Measure: Number; unit: participants
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
participants
  Less Than | 1
  More Than | 0
  Equal to | 3

4. Primary Outcome: Requirement for Blood Transfusion
Description: Number of blood transfusions required (units of packed red blood cells or units of whole blood) or infusion of autologous red cells during and after surgery
Time Frame: during and after surgery
Population: as for outcome 1
Measure: Number; unit: number of transfusions
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
number of transfusions | 0

5. Primary Outcome: Number of Post Operative Bleeding Episodes (See Table Below)
Description: Bleeding was assessed at least once each day by the investigator, more frequently if indicated by the severity of the operation or the subject's response. This included all bleeding episodes from the end of the surgical procedure until the subject was no longer at risk of bleeding due to surgery
Time Frame: End of surgery till end of study
Population: as for outcome 1
Measure: Number; unit: number of bleeds
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
number of bleeds | 0

6. Primary Outcome: Change of Haemoglobin From Pre-surgery Till End of Treatment
Description: The subject's haemoglobin was measured pre operatively, within 2 hours post operatively and at the End of Treatment Assessment. Changes in the subject's haemoglobin from pre to post operatively and from post operatively to the End of Treatment Assessment were assessed, taking into account the volume of fluid infused into the subject during the intervening periods, any blood transfusions in the intervening periods, the subject's haematocrit at the same time points and the subject's pre dose serum ferritin
Time Frame: 2 hrs pre-operatively till end of treatment
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: g/L
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
g/L | -36.0 (26.17)

7. Secondary Outcome: Dose Per Infusion (IU/kg)
Description: weight adjusted dose per infusion until a subject was no longer at risk of bleeding due to surgery
Time Frame: before surgery, during the post operative period
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/kg
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
IU/kg | 16.14 [10.13 to 22.30]

8. Primary Outcome: Number of Participants With Degree of Bleeding Control Rated as Excellent.
Description: Investigators made an overall assessment of FACTOR X in controlling bleeding at the End of Treatment Assessment. The degree of bleeding control was rated as excellent, good, poor or unassessable, in accordance with the following criteria listed below:
  * Excellent -Parameters were similar to those in subjects without a bleeding disorder.
  * Good -Parameters were inferior to those in subjects without a bleeding disorder, but no other factor X containing agents were required to restore haemostasis.
  * Poor - Blood loss was excessive (defined as more than twice the pre defined amount that would be expected in a subject without a bleeding disorder for this type of surgery) and/or Haemostasis was not achieved and/or Additional factor X containing agents were required to restore haemostasis.
  * Unassessable -Efficacy was not possible to assess, or Additional factor X containing agents (excluding blood transfusions) were required before efficacy of FACTOR X could be assessed.
Time Frame: During and till end of treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Active Treatment With FACTOR X
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the date the Informed Consent Form was signed until the end of the subject's participation in the study
Description: Treatment-emergent AEs are defined as AEs occurring or worsening after the start (date and time) of the first study treatment until End of Treatment Assessment or follow-up safety assessment (28 days after the last dose of FACTOR X) if performed
Arm/Group | FACTOR X
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FACTOR X (N=4)
Haematoma (Vascular disorders) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Procedural pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
none reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days